CLINICAL TRIAL: NCT03397355
Title: Changes of Tumor-related Biomarkers Before and After Pulmonary Nodule Biopsy and Their Clinical Implications.
Brief Title: Monitoring the Changes of Tumor-related Biomarkers Before and After Pulmonary Nodule Biopsy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Chen Wang, Professor, China-Japan Friendship Hospital
Other Study IDs: Lung biopsy and biomarkers
Record Dates: First submitted 2017-12-30; First posted 2018-01-12 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: Pulmonary Nodule; Lung Cancer; Biopsy; Biomarker.
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the past few years, circulating tumor cells (CTCs), circulating tumor DNA (ctDNA), microRNAs, autoantibodies, and T-cell receptor repertoire are new biomarkers of liquid biopsy in cancer, which has been demonstrated to have a great value in diagnostics, treatment evaluation, and prognosis prediction. However, most of previous data were based on late stage tumor patients. This study plans to utilize the minimally invasive method to detect the changes of numbers of CTCs, ctDNA hot spot mutations and methylation signals, microRNAs, autoantibodies, and T-cell receptor repertoire in early stage lung cancer patients before and after pulmonary nodule biopsy, during therapeutic and follow-up periods, in order to evaluate the clinical values of above tumor-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as suspected lung cancer patients with pulmonary nodules (single or multiple) by CT scans, and the maximum diameter of nodule is between 8mm and 3cm;
* Male or female, with age of 18~80 years;
* Agree to take the pulmonary nodule biopsy, and sign the Informed Consent.

Exclusion Criteria:

* With severe comorbidities and unable to participate in this study;
* Diagnosed with acute respiratory tract infection, for instance fungus, mycobacterium tuberculosis or other bacteria, virus, etc., one month prior to the study recruitment;
* Pregnant or maternal women;
* Diagnosed with other carcinoma, and the pulmonary nodules suspected of stemming from other sites;
* Unable for regular follow-ups according to the research protocol;
* Blood sample is not qualified for biomarker testing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodules (single or multiple) by CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Death or survival | Baseline and every three- or six-month follow-up within two years for each patient.
  Death or survival
Disease progress | Baseline and every three- or six-month follow-up within two years for each patient.
  Complete Response(CR), Partial Response(PR), Stable Disease(SD), Progressive Disease(PD)
Reasons of study termination | Baseline and every three- or six-month follow-up within two years for each patient.
  Complete the study, Lost to follow-up, Withdrawal of informed consent, Terminated by the investigator, Severe adverse event(SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Chen WANG, Ph.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China